CLINICAL TRIAL: NCT06043531
Title: Targeting Trimethylamine N-Oxide for Cardiovascular Health In Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20027920
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVOO supplementation (Experimental): 50g/day, dietary supplementation Extra Virgin Olive Oil (EVOO)
  Interventions: Other: Experimental: EVOO
- Standard of Care (No Intervention): Standard of care control

INTERVENTIONS:
Other: Experimental: EVOO — Subjects will consume 50g of cold pressed EVOO per day for 28 days.
  Other Names: Dietary EVOO
  Arms: EVOO supplementation

SUMMARY:
Despite medical and surgical advances, long-term survival in liver transplant (LT) recipients is compromised by an increased risk of cardiovascular disease (CVD) after transplant, the mechanisms of which are still not fully understood. TMAO is an attractive therapeutic target to improve vascular health and diastolic function toward preventing CVD in LT patients. Therefore, the purpose of this study is to better understand the role of TMAO in cardiovascular dysfunction patients with chronic kidney disease.

DETAILED DESCRIPTION:
Despite medical and surgical advances, long-term survival in liver transplant (LT) recipients is compromised by an increased risk of cardiovascular disease (CVD) after transplant, the mechanisms of which are still not fully understood. Following LT, patients have an increased incidence of atherosclerotic CVD. Notably, atherosclerotic CVD is an established risk factor for diastolic dysfunction and incident heart failure with preserved ejection fraction (HFpEF). There is a critical need to better understand the biological mechanisms of LT related vascular dysfunction and establish targeted interventions that will reduce the risk of CVD in this patient population. In the general population, there is strong epidemiological evidence linking high TMAO levels with atherosclerotic CVD and heart failure, and that it can modulated rapidly by diet within two weeks. Therefore, the purpose of this study is to better understand the role of TMAO in cardiovascular dysfunction patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Speak and understand English
* Have received and LT

Exclusion Criteria:

* Acute cellular or chronic rejection within 3 months
* Post-LT liver or non-liver related malignancy
* Active viral hepatitis (B or C) or autoimmune hepatitis
* Untreated biliary strictures or vascular complications (e.g. hepatic artery thrombosis)
* Poorly controlled diabetes (HbA1c >8.5%)
* Relapse of alcohol use after LT
* Follow a vegetarian or vegan diet
* Current pregnancy
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Serum TMAO | Change from baseline at four weeks
  Serum TMAO levels will be assessed by nuclear magnetic resonance (NMR)

SECONDARY OUTCOMES:
Conduit artery endothelial function changes | Change from baseline at four weeks
  Conduit artery endothelial function assessed by flow mediated dilation
Microvascular function change | Change from baseline at four weeks
  Skin blood flow response to local heating measured by laser doppler flowmetry
Arterial hemodynamics changes | Change from baseline at four weeks
  Arterial hemodynamics derived from radial artery tonometry recordings
Diastolic Function change | Change from baseline at four weeks
  Diastolic function at rest by echocardiography and during isometric handgrip exercise
Frailty outcome hanges | Change from baseline at four weeks
  Frailty outcomes assessed according to Fried criteria
Quality of life changes | Change from baseline at four weeks
  Quality of Life assessed by SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kirkman, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States